CLINICAL TRIAL: NCT02288442
Title: Exercise Training (WHOLEi+12) in Pulmonary Hypertension
Brief Title: Whole Muscle Exercise Training (WHOLEi+12) in Pulmonary Hypertension
Acronym: WHOLEi+12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alejandro Lucia, Prof, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEMadrid
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Exercise Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention)
- exercise (Experimental): exercise intervention during 8 weeks
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Exercise training for 8 weeks (aerobic exercise, resistance training and inspiratory muscle training thrice a week)
  Arms: exercise

SUMMARY:
The purpose of this RCT is to study the effects of whole muscle training (inspiratory muscle training + aerobic training + muscle resistance training) on muscle power, VO2peak and gas-exchange variables obtained during cardiopulmonary exercise testing, QoL, functional capacity (eg, 6-min walking distance), and maximal inspiratory pressure in patients with pulmonary artery hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed pulmonary hypertension, class II-III NYHA, no syncope in the last 3 months (stable clinical condition) or chronic thromboembolic pulmonary hypertension

Exclusion Criteria:

* Not meeting the above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Muscle power (upper and lower-body) | 8 weeks

SECONDARY OUTCOMES:
6 minute walk distance test | 8 weeks
maximal inspiratory pressure (PImax) | 8 weeks
Short Form 36-Item Health Survey questionnaire version 2 (SF-36) | 8 weeks
Physical activity levels objectively determined with accelerometry | 8 weeks
Peak oxygen uptake (VO2peak) directly measured during cardiopulmonary exercise testing (CEPT) | 8 weeks
Other CEPT variables | 8 weeks
  Gas-exchange variables at the anaerobic threshold
NT-ProBNP | 8 weeks
Performance in the 5-repetition sit-stand-test (5SST) | 8 weeks
Safety assessment | 8 weeks
  Evaluation of adverse episodes, ie. syncopal/pre-syncopal episodes, severe dyspnea, arrhythmias, asthma, signs of poor peripheral perfusion or central nervous symptoms (ataxia, tremors). These episodes were be reported directly by the study researchers (in the exercise group) and by a telephone interview every 2 weeks in all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 12 de Octubre, Madrid, Madrid, Spain